CLINICAL TRIAL: NCT06975878
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, 2-arm Study to Investigate the Safety and Immunogenicity of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers
Brief Title: Study of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants From Approximately 2 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK04; 2023-507600-32 (Registry Identifier: CTIS); U1111-1295-6064 (Other: WHO ICTRP)
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Immunization; Healthy Volunteers
MeSH Terms: interventions — DTaP-IPV-HB-PRP-T vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind
  * Blinding for vaccine group assignment: participants and participant's parent(s) / legally acceptable representative(s) (LARs), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: those preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 2-dose primary series of PCV21 at approximately 2 and 4 months of age (MoA) or a 3-dose primary series (preterm infants) at 2, 3, and 4 MoA co- administered with Hexyon. At 11 to 15 MoA, participants will receive a 3rd dose or 4th dose (for preterm infants) of PCV21 co-administered with Hexyon and M M RvaxPro; Varivax will also be co-administered unless not possible as per local practice
  Interventions: Biological: PCV21 vaccine; Biological: Hexyon vaccine; Biological: M-M-RvaxPro vaccine; Biological: Varivax vaccine
- Group 2: 15vPCV (Active Comparator): Participants will be administered via intramuscular injection (IM) a 2-dose primary series of 15vPCV at approximately 2 and 4 months of age (MoA) or a 3-dose primary series (preterm infants) at 2, 3, and 4 MoA co- administered with Hexyon. At 11 to 15 MoA, participants will receive a 3rd dose or 4th dose (for preterm infants) of 15vPCV co-administered with Hexyon and M M RvaxPro; Varivax will also be co-administered unless not possible as per local practice
  Interventions: Biological: Vaxneuvance vaccine; Biological: Hexyon vaccine; Biological: M-M-RvaxPro vaccine; Biological: Varivax vaccine

INTERVENTIONS:
Biological: PCV21 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: 515
  Arms: Group 1: PCV21
Biological: Vaxneuvance vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Vaxneuvance ™
  Arms: Group 2: 15vPCV
Biological: Hexyon vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Hexyon®
Biological: M-M-RvaxPro vaccine — Pharmaceutical form:Powder and solvent for suspension for injection-Route of administration:Intramuscular or Subcutaneous
  Other Names: M-M-RVAX-PRO®
Biological: Varivax vaccine — Pharmaceutical form:Powder and solvent for suspension for injection-Route of administration:Intramuscular or Subcutaneous
  Other Names: Varivax®

SUMMARY:
This study is a Phase 3, randomized, modified double-blind study which aims to measure whether PCV21 vaccine (investigational pneumococcal conjugate vaccine) is safe and can help the body to develop germ-fighting agents called "antibodies" (immunogenicity) compared with 15vPCV (Vaxneuvance, licensed pneumococcal conjugate vaccine) when they are administered with routine pediatric vaccines in infants aged from approximately 2 months (42 to 112 days).

The study duration per participant will be up to approximately 20 months. The study vaccines (either PCV21 or 15-valent pneumococcal vaccines) will be administered at approximately 2, 4, and 11 to 15 months of age or at approximately 2, 3, 4, and 11 to 15 months of age (for preterm infants). Routine pediatric vaccines will be given at the same timepoints, as per local practice / recommendations.

• There will be 5 (for full-term infants) or 6 (for preterm infants) study visits:

* Full-term infants: Visit (V)01, V02 separated from V01 by 60 days, V03 separated from V02 by 30 days, V04 at 11 months of age until 15 months of age, V05 separated from V04 by 30 days.
* Preterm infants: Visit (V)01, V02 separated from V01 by 30 days, V03 separated from V02 by 30 days, V04 separated from V03 by 30 days, V05 at 11 months of age until 15 months of age, V06 separated from V05 by 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 112 days on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable as assessed by the investigator

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed Streptococcus pneumoniae infection or disease
* Any contraindication to the routine pediatric vaccines being administered in the study
* History of seizure or significant stable or progressive neurological disorders such as infantile spasms, inflammatory nervous system diseases, encephalopathy, cerebral palsy
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Laboratory-confirmed or known thrombocytopenia, as reported by the parent/legally acceptable representative (LAR), contraindicating intramuscular (IM) injection
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 4 weeks following the study intervention administration, except for oral rotavirus vaccine, which may be received anytime during the study including at study visits and for influenza vaccination or meningococcal b vaccine, which may be received at least 14 days before or 14 days after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines, as applicable per local recommendations.
* Previous vaccination against S. pneumoniae
* Previous vaccination against the following antigens: diphtheria, tetanus, pertussis, Haemophilus influenzae type b, and poliovirus
* Receipt of more than 1 dose of hepatitis B vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 42 Days to 112 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1080 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Seroresponse rate for PCV21 and 15vPCV serotypes | 30 days post-toddler dose
  Serotype specific IgG concentration ≥ 0.35 µg/mL
IgG concentration for PCV21 and 15vPCV serotypes | 30 days post-toddler dose
  Serotype specific IgG Geometric Mean Concentration (GMC)

SECONDARY OUTCOMES:
Anti- hepatitis B surface antigen (HBsAg) Ab | 30 days post-toddler dose
  % Antibody concentrations ≥ 10 milli international units per milliliter (mIU/mL)
Anti- polyribosylribitol phosphate (PRP) Ab | 30 days post-toddler dose
  % Antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL)
Anti-poliovirus types (1, 2, and 3) Ab | 30 days post-toddler dose
  % Antibody titers ≥ 1:8
Anti-diphtheria Ab concentrations | 30 days post-toddler dose
  % Antibody concentration ≥ 0.1 IU/mL
Anti-tetanus Ab concentrations | 30 days post-toddler dose
  % Antibody concentration ≥ 0.1 IU/mL
Anti-pertussis Ab concentrations (Pertussis toxin (PT) and Filamentous Hemagglutinin (FHA)) | 30 days post-toddler dose
  Antibody GMC
Anti-measles Ab concentrations | 30 days post-toddler dose
  Antibody GMC
Anti-mumps Ab concentrations | 30 days post-toddler dose
  Antibody GMC
Anti-rubella Ab concentrations | 30 days post-toddler dose
  Antibody GMC
Anti-varicella Ab concentrations | 30 days post-toddler dose
  Antibody GMC
Anti HBsAg concentrations | 30 days post-primary series
  % Antibody concentrations ≥ 10 mIU/mL
Anti-PRP Ab concentrations | 30 days post-primary series
  % Antibody concentrations ≥ 0.15 µg/mL
Anti-poliovirus types (1, 2, and 3) Ab titers | 30 days post-primary series
  % Antibody titers ≥ 1:8
Anti-diphtheria Ab concentrations | 30 days post-primary series
  % Antibody concentrations ≥ 0.1 IU/mL
Anti-tetanus Ab concentrations | 30 days post-primary series
  % Antibody concentrations ≥ 0.1 IU/mL
Anti-pertussis Ab concentrations (PT and FHA) | 30 days post-primary series
  Antibody GMC
Serotype specific OPA titers for all serotypes included in PCV21 | 30 days post-primary series
  Antibody Geometric mean titer (GMT)
Serotype specific OPA titers for all serotypes included in PCV21 | 30 days post-toddler dose
  Antibody GMT
Presence of any immediate adverse events (AEs) | Within 30 minutes after each vaccine injection
  Number of participants experiencing immediate AEs
Presence of solicited injection site and systemic reactions through 7 days after each vaccine injection | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site and systemic reactions
Presence of unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs through 30 days after each vaccine injection | Through 30 days after each vaccine injection
  Number of participants experiencing unsolicited injection site reactions and unsolicited systemic AEs
Presence of serious adverse events (SAEs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 20 months
  Number of participants experiencing SAEs
Presence adverse events of special interest (AESIs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 20 months
  Number of participants experiencing AESIs

CONTACTS AND LOCATIONS:
Locations (48):
- Belgium (6):
  - Investigational Site Number : 0560004, Alken
  - Investigational Site Number : 0560001, Bruges
  - Investigational Site Number : 0560002, Edegem
  - Investigational Site Number : 0560005, Gozée
  - Investigational Site Number : 0560007, Leuven
  - Investigational Site Number : 0560003, Roeselare
- Czechia (4):
  - Investigational Site Number : 2030001, Jindřichův Hradec
  - Investigational Site Number : 2030009, Krnov
  - Investigational Site Number : 2030006, Pilsen
  - Investigational Site Number : 2030008, Prague
- Estonia (3):
  - Investigational Site Number : 2330001, Paide
  - Investigational Site Number : 2330004, Tallinn
  - Investigational Site Number : 2330002, Tartu
- Finland (9):
  - Investigational Site Number : 2460008, Espoo
  - Investigational Site Number : 2460001, Helsinki
  - Investigational Site Number : 2460010, Helsinki
  - Investigational Site Number : 2460005, Jarvenpaa
  - Investigational Site Number : 2460003, Kokkola
  - Investigational Site Number : 2460004, Oulu
  - Investigational Site Number : 2460002, Seinäjoki
  - Investigational Site Number : 2460007, Tampere
  - Investigational Site Number : 2460009, Turku
- Germany (8):
  - Investigational Site Number : 2760005, Herxheim
  - Investigational Site Number : 2760006, Hürth
  - Investigational Site Number : 2760014, Hürth
  - Investigational Site Number : 2760013, Krefeld
  - Investigational Site Number : 2760010, Mönchengladbach
  - Investigational Site Number : 2760012, Mönchengladbach
  - Investigational Site Number : 2760008, Schönau am Königssee
  - Investigational Site Number : 2760003, Wolfsburg
- Greece (3):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000006, Ioannina
  - Investigational Site Number : 3000005, Thessaloniki
- Italy (7):
  - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800004, Rome, Roma
  - Investigational Site Number : 3800001, Bari
  - Investigational Site Number : 3800008, Foggia
  - Investigational Site Number : 3800010, Lecce
  - Investigational Site Number : 3800007, Milan
  - Investigational Site Number : 3800009, Parma
- Poland (8):
  - Investigational Site Number : 6160001, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160007, Torun, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160009, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160003, Trzebnica, Lower Silesian Voivodeship
  - Investigational Site Number : 6160008, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160005, Dziekanów Leśny, Masovian Voivodeship
  - Investigational Site Number : 6160011, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160002, Siemianowice Śląskie, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PSK04 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26678&tenant=MT_SNY_9011